CLINICAL TRIAL: NCT05752526
Title: A Phase 1, Multi-site, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Pharmacokinetics, Safety and Preliminary Efficacy of Two Strengths of DARE-PDM1 (1% or 3%) Versus Placebo Among Women With Symptomatic Primary Dysmenorrhea
Brief Title: A Study of Diclofenac Gel in Women With Primary Dysmenorrhea
Acronym: DARE-PDM1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DARE-PDM1-001
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Dysmenorrhea Primary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DARE-PDM1 1% Diclofenac Vaginal Gel (Experimental): 1% Diclofenac in 2.5 mL Hydrogel
  Interventions: Drug: Diclofenac 1%
- DARE-PDM1 3% Diclofenac Vaginal Gel (Experimental): 3% Diclofenac in 2.5 mL Hydrogel
  Interventions: Drug: Diclofenac 3%
- Placebo (Placebo Comparator): 2.5 mL Hydrogel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac 1% — vaginal hydrogel containing 1% Diclofenac
  Arms: DARE-PDM1 1% Diclofenac Vaginal Gel
Drug: Diclofenac 3% — vaginal hydrogel containing 3% Diclofenac
  Arms: DARE-PDM1 3% Diclofenac Vaginal Gel
Drug: Placebo — vaginal hydrogel, no active ingredient
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare 1% and 3% diclofenac gel (DARE-PDM1) to placebo in women with symptomatic primary dysmenorrhea. The main question it aims to answer are:

Is DARE-PDM1 1%, 3% diclofenac gel systemically safe? What are the systemic levels of DARE-PDM1 1%, 3% diclofenac gel in plasma and vaginal fluid following 1 dose and 3 doses.

Participants will be seen for routine safety evaluations and complete a daily diary recording dysmenorrhea associated pain.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18- 50 years old (inclusive)
* Self-assessment of historic dysmenorrhea associated pain level of ≥ 5 on a scale of 0 - 10 in at least one of the following anatomic sites: pelvic/vaginal pain, low back pain, while not using NSAIDs or hormonal contraception.
* Non-pregnant status
* If applicable, agrees to be sexually abstinent and place nothing in the vagina during the 120 hours between visits 3 and 8 and the 3-day period of the multiple dose regimen.
* Agrees to use adequate non-hormonal birth control during the trial (e.g. study provided male condoms without nonoxynol-9 lubricant, tubal sterilization, heterosexual abstinence) (Because hormonal birth control is a known off label treatment for dysmenorrhea, if the participant is on hormonal birth control other than Depo-Provera contraceptive injection, she agrees to discontinue it and have at least one spontaneous intervening menses before the start of the study period. If using Depo Provera, has not had an injection within the 4 months before Visit 1 and must have had a spontaneous menses prior to visit 2.)
* Provides informed consent for participating in the trial
* Willingness to use only study-provided oral paracetamol as rescue pain medication for dysmenorrhea, if needed according to investigator's instruction.
* Patient is fluent in the English language.
* Patient is capable of understanding and complying with the protocol and agrees to sign the informed consent document.
* Patient has had a cervical screen performed within five years prior to Visit 1 and can provide documentation indicating normal test results consistent with Australian Health guidelines. If the patient cannot provide documentation, a cervical screen will be performed at Visit 1. Patients with abnormal findings will be excluded from study participation and be referred for follow-up medical care as appropriate.

Exclusion Criteria:

* Positive pregnancy test
* Unwilling or unable to comply with protocol
* Allergic to diclofenac or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients with severe liver, kidney or heart failure
* After the use of aspirin or other nonsteroidal anti-inflammatory drugs, asthma, nasal polyps, angioedema and urticaria have occurred in the past
* Current active peptic ulcer bleeding or perforation
* Have a history of significant upper gastrointestinal disease
* Have a chronic pain syndrome other than dysmenorrhea which could confound preliminary efficacy data (e.g., chronic low back pain unrelated to menses)
* Have a positive Sexually Transmitted Infection (STI) test at screening for Chlamydia trachomatis or Neisseria gonorrhea

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Measure the systemic Level of Diclofenac after a single dose of DARE-PDM1 | 7 days
  Evaluate the plasma pharmacokinetics of diclofenac after a single dose of DARE-PDM1
Measure the systemic Level of Diclofenac after three doses of DARE-PDM1 | 3 days
  Evaluate the plasma pharmacokinetics of diclofenac after three doses of DARE-PDM1
Measure the Vaginal Fluid levels of diclofenac after three doses of DARE-PDM1 | 3 days
  Evaluate the vaginal fluid pharmacokinetics of diclofenac after three doses of DARE-PDM1
Measure the Vaginal Fluid levels of diclofenac after a single dose DARE-PDM1 | 7 days
  Evaluate the vaginal fluid pharmacokinetics of diclofenac after a single dose of DARE-PDM1
Number of participants with abnormal vaginal exam findings. | 60 days
  Compare genital safety of DARE-PDM1 versus placebo through vaginal exams
Number of participants with abnormal laboratory test results. | 60 days
  Evaluate systemic safety of DARE-PDM1 versus placebo through safety laboratory assessments

OTHER OUTCOMES:
Number of participants that record a decrease in dysmenorrhea associated pain | 60 days
  Evaluate the efficacy of DARE-PDM1 versus placebo in reducing dysmenorrhea associated pain
Use of Rescue Medications | 60 days
  Evaluate the number of pain medication doses needed while using DARE-PDM1

CONTACTS AND LOCATIONS:
Locations (1):
- PARC Clinical Research, Adelaide, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
A decision has not yet been made on when or what IPD to share when available.